CLINICAL TRIAL: NCT03150316
Title: A Phase I, Open-Label, Multi-Center Study of CKD-581 in Combination With Lenalidomide and Dexamethasone in Patients With Previously Treated Multiple Myeloma
Brief Title: CKD-581 + Lenalidomide + Dexamethasone in Patients With Previously Treated Multiple Myeloma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 133MM16016
Record Dates: First submitted 2017-05-10; First posted 2017-05-12 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Myeloma, Multiple
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treat Regimen (Experimental): CKD-581(investigational Drug) Lenalidomide Dexamethasone
  Interventions: Drug: Treat Regimen

INTERVENTIONS:
Drug: Treat Regimen — CKD-581(investigational Drug): on days 1, 8, 15 of repeated 28day cycles Lenalidomide: on days 1~21 of repeated 28 day cycles Dexamethasone: administrated once weekly every 28day cycles
  Other Names: CKD-581 lenalidomide dexamethasone regimen

SUMMARY:
This study is to determine the maximum tolerated dose(MTD) and recommened phase 2 dose(RP2D) based on dose limiting toxicity(DLT), and to evaluate safety and pharmacokinetics(PK) profile of a single agent CKD-581 injection in Combination with Lenalidomide and Dexamethasone in patients with Previously Treated Multiple Myeloma.

DETAILED DESCRIPTION:
This is an open label, dose escalation study. Cohort of 3~6 patients receive escalation doses of CKD-516 until the maximum tolerated dose(MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

* must have received at least two prior lines of therapy and Diagnosis of symptomatic multiple myeloma(IMWG 2015)
* Eastern Cooperative Oncology Group performance status ≤ 2
* Life expectancy 12 weeks
* must have the following laboratory values within 3 weeks prior to first dose of study drug

  * absolute neutrophil count(ANC) ≥ 1,500 mm3
  * platelet count(PLT)≥ 100,000 mm3
  * Hb ≥ 9.0g/dL
  * AST(SGOT) and ALT(SGPT) ≤ 3 x upper limit of normal(UNL)
  * Serum bilirubin ≤ 1.5 x ULN (but, Gilbert syndrome ≤ 3 x UNL)
  * Creatinin Clearance(CrCl) ≤ 50mL/min
* One more measureable disease following values

  * Serum M-protein ≥ 1g/dL
  * Urine M-Protein ≥ 200mg/24hr
  * in that case serum M-protein, urine M-Protein nonmeasurable and FLC ratio abnormal, Serum free light chain(FLC) level ≥ 100mg/L(≥10mg/dL)
* more than 24 weeks prior to last lenalidomide dose
* must have signed the consent form

Exclusion Criteria:

* Patients with CNS disease
* Patients with clinically significant heart disease within 24weeks prior to first dose of study drug
* patients with clinically significans abnormal EKG, echocardiography at screening
* patients with patients with embolism within 24 weeks
* patients with active hepatitis, HIV positive(exception, non active hepatitis)
* peripheral neuropathy ≥ CTCAE grade 2 within 2 weeks prior to first dose of study drug
* Patients with clinically significant disease
* Patients with a prior malignancy with in the last 3 years except adequately treated basal cell or squamous cell or skin cancer, in situ cervical cancer
* Patients who have received surgery, chemotherapy, radiation therapy or immunotherapy or any other investigational drugs ≤ 4 weeks prior to first dose of study drug and during treatment period
* Patients who can not anticoagulate
* Patients who have received dexamethasone >10mg/day within 2week prior to first dose of study drug and during treatment period
* Women who are pregnant or breast feeding or women of childbearing potential not using an effective method of birth control. Male patients whose sexual partners are not using effective birth control.
* patients with hypersensitive reaction of lenalidomide or dexamethasone

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
MTD | Up to 28 days(for 1st cycle)
  Maximum Tolerated Dose

SECONDARY OUTCOMES:
Pharmacokinetics(Cmax) | 1st Cycle day1: up to 24hr
  Pharmacokinetics

OTHER OUTCOMES:
Objective Response Rate(ORR) | Average time period between the start day of induction therapy and the day of relapse or progression or death, whichever occurs firstly, up to 1year
  Objective Response Rate(ORR) of participants as assessed by IMWG uniform response criteria(2011) every 4weeks
Progression Free Survival(PFS) | Average time period between the start day of induction therapy and the day of relapse or progression or death, whichever occurs firstly, up to 1year
  Progression Free Survival(PFS) of participants as assessed by IMWG uniform response criteria(2011) every 4weeks
Overall Survival(OS) | Average time period between the start day of induction therapy and the day of death, due to any cause, up to 1year
  Overall Survival(OS) of participants as assessed by IMWG uniform response criteria(2011) every 4weeks
Duration of Response(DOR) | Average time period between the day of first achievement of response and the day of first relapse or progression, up to 1year
  Duration of Response(DOR) of participants as assessed by IMWG uniform response criteria(2011) every 4weeks
Pharmacokinetics(T1/2) | 1st Cycle day1: up to 24hr
  Pharmacokinetics
Pharmacokinetics(CL) | 1st Cycle day1: up to 24hr
  Pharmacokinetics
Pharmacokinetics(AUClast) | 1st Cycle day1: up to 24hr
  Pharmacokinetics
Pharmacokinetics(AUCinf) | 1st Cycle day1: up to 24hr
  Pharmacokinetics
Pharmacokinetics(Vd) | 1st Cycle day1: up to 24hr
  Pharmacokinetics
Pharmacokinetics( MRT) | 1st Cycle day1: up to 24hr
  Pharmacokinetics
Adverse events | through study completion, an average of 1 year
  Adverse events will be assessed using CTCAE criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Chanki Min, Principal Investigator — The Catholic University of Korea
Locations (2):
- South Korea (2):
  - Samsung Hospital, Seoul, Gangnam-gu
  - the catholic university of korea, Seoul ST. Mary's Hospital, Seoul, Seocho

IPD SHARING:
Plan to Share IPD: No